CLINICAL TRIAL: NCT01884909
Title: An Open Label, Randomized, Two-Period, Two-Treatment, Two-Sequence, Crossover, Balanced, Single Dose Oral Bioequivalence Study of Metoprolol Succinate Extended Release Tablets 200 mg of Ipca Laboratories Limited, India and 'Toprol-XL®' (Metoprolol Succinate) Extended Release Tablets 200 mg of Astrazeneca LP, USA In Healthy Adult Human Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Metoprolol Succinate Extended Release Tablets 200 mg Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA1264351
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 'TOPROL-XL®' ER Tablets 200 mg (Active Comparator): 'TOPROL-XL®' ER Tablets 200 mg of Astrazeneca LP, USA
  Interventions: Drug: Metoprolol Succinate ER Tablet 200 mg; Drug: 'TOPROL-XL®' ER Tablets 200 mg
- Metoprolol Succinate ER Tablet 200 mg (Experimental): Metoprolol Succinate ER Tablet 200 mg of Ipca Laboratories Limited, India
  Interventions: Drug: Metoprolol Succinate ER Tablet 200 mg; Drug: 'TOPROL-XL®' ER Tablets 200 mg

INTERVENTIONS:
Drug: Metoprolol Succinate ER Tablet 200 mg — 1 * 200 mg tablet per day
  Other Names: Test product
Drug: 'TOPROL-XL®' ER Tablets 200 mg — 1 * 200 mg tablet per day
  Other Names: Reference product

SUMMARY:
This is an open Label, randomized, two-period, two-treatment, two-sequence, crossover, balanced, single dose pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fed condition in healthy adult human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Metoprolol Succinate 200 mg Ipca Laboratories Limited, India and the corresponding Reference Product: TOPROL-XL® (Metoprolol Succinate) extended release Tablets 200 mg of Astrazenica LP, USA under fed condition in healthy adult human subjects in a randomized crossover study.

The study was conducted with 48 healthy adult subjects. In each study period, a single 200 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was approximately 11 days including washout period of at least 7 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years old, both inclusive.
2. Sex: Males and/or non-pregnant, non-lactating females.
3. BMI: 18.5 to 24.9 weight in kg/(height in meter)2 both inclusive;
4. Able to communicate effectively with study personnel and willingness to follow the protocol requirements as evidenced by written informed consent.
5. Able to give written informed consent to participate in the study.
6. All volunteers must be judged by the principal or co-investigator or physician as normal and healthy during a pre-study safety assessment performed within 21 days of the first dose of study medication which will include:

   * A physical examination with no clinically significant finding.
   * Results within normal limits or clinically non-significant for the tests mentioned in List of Laboratory Parameters:
   * Additional tests and/or examinations may be performed, if necessary, based on Principal Investigator discretion.
   * All results will be assessed against the laboratory normal ranges current at the time of testing and a copy of the normal ranges used will be included in the study documentation.

Exclusion Criteria:

1. History of allergic responses to Metoprolol Succinate or other related drugs, or any of its formulation ingredients.
2. Have significant diseases or clinically significant abnormal findings during screening, [medical history, physical examination, laboratory evaluations, ECG, chest X-ray recording, obstetrics and gynecological history and examination along with PAP smear (for female volunteers) & transvaginal ultrasonography (for female volunteers)].
3. Any disease or condition which might compromise the haemopoeitic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
4. History or presence of bronchial asthma.
5. Use of any hormone replacement therapy within 3 months prior to study medication dosing.
6. A depot injection or implant of any drug within 3 months prior to administration of study medication.
7. Use of enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
8. History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
9. Smokers who smoke 10 or more cigarettes per day or 20 or more biddies per day or those who cannot refrain from smoking during the study period.
10. History of difficulty with donating blood or difficulty in accessibility of veins.
11. History of allergic response to heparin.
12. A positive hepatitis screen (includes subtypes B & C).
13. A positive test result for HIV antibody and / or syphilis (RPR/VDRL).
14. Volunteers who have donated blood (1 unit or 450 mL) within 90 days prior to the initial dose of the study drug or have blood loss, excluding volume drawn at screening for this study, (≤100 mL within 30 days; ≤200 mL within 60 days; >200 mL within 90 days) prior to initial dose of study drug.
15. History of difficulty in swallowing, or of any gastrointestinal disease which could affect drug absorption.
16. Intolerance to venipuncture
17. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Co-Investigator, could contraindicate the volunteer's participation in this study.
18. Volunteers who have received a known investigational drug within five elimination half life of the administered drug prior to the initial dose of study drug or who have participated in a clinical drug study or bioequivalence study within 90 days prior to the initial dose of study drug, whichever is greater.
19. Found positive in urine test for drugs of abuse done before check-in of period I.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 1 Month
  Area Under Curve (AUC)and Cmax Sampling Hours: Pre-dose and at 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0,11.0, 12.0, 13.0, 14.0, 16.0, 20.0, 24.0, 36.0 and 48.0 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Manish Singhal, M.B.B.S, Principal Investigator — Cliantha Research Limited
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India